CLINICAL TRIAL: NCT06657625
Title: Impact of the Introduction of a Performance Improvement Program on the Initial Management of Sepsis and Septic Shock in Adults in the Emergency Department: a Before-and-after Study
Brief Title: Impact of the Introduction of a Performance Improvement Program on the Initial Management of Sepsis and Septic Shock in Adults in the Emergency Department: a Before-and-after Study (IPA-SOS)
Acronym: IPA-SOS
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0223 - IPA-SOS
Record Dates: First submitted 2024-10-14; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-07

CONDITIONS: Sepsis; Septic Shock; Critical Illness; Emergency Medicine; Surviving Sepsis Campaign; Sepsis Performance Improvement Program; Sepsis Team
MeSH Terms: conditions — Sepsis; Shock, Septic; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-implementation cohort: Patients from January 1, 2017, to December 31, 2017, before the implementation of the performance improvement program.
- Post-implementation cohort: Patients from May 1, 2022, to April 30, 2024, after the implementation of the performance improvement program.
  Interventions: Other: Sepsis Performance Improvement Program

INTERVENTIONS:
Other: Sepsis Performance Improvement Program — Training/awareness for medical and paramedical staff; creation of informational posters; development of an institutional pathway in the emergency department; creation of a protocol ; establishment of a sepsis team with a dedicated contact number.
  Other Names: Implementation of a Performance Improvement Program; Performance Improvement Program
  Groups: Post-implementation cohort

SUMMARY:
The goal of this observational study is to evaluate if a performance improvement program can improve the initial management of sepsis and septic shock in adults at Brest University Hospital. The study will include adult patients with positive blood cultures and a positive SOFA (Sequential Organ Failure Essessment) score, or with blood cultures collected, a positive SOFA score, and sepsis/septic shock confirmed by the sepsis team at Brest University Hospital.

The main questions it aims to answer are:

* Does the implementation of a performance improvement program increase adherence to the 2021 Surviving Sepsis Campaign (SSC) guidelines?
* Does the program improve patient outcomes, such as 90-day mortality, progression to septic shock, and length of stay in the ICU and hospital?

Researchers will compare patients from two periods : pre-implementation (January 1, 2017 to December 31, 2017) and post-implementation (May 1, 2022 to April 30, 2024), to see if the performance improvement program leads to better compliance with SSC guidelines and improved patient outcomes.

Participants will:

* Have their clinical data (such as blood cultures, SOFA scores, and treatment times) collected and analyzed.
* Be monitored for time to antibiotic therapy, initial fluid resuscitation, and other key treatment interventions following the recognition of sepsis or septic shock.

DETAILED DESCRIPTION:
Sepsis and septic shock are conditions with a significant public health impact, yet the incidence of sepsis continues to rise. To improve the management of these conditions, experts recommend implementing performance improvement programs. These recommendations were applied at Brest University Hospital in 2018, including the creation of a "sepsis team" responsible for prevention, education, and providing guidance and advice on sepsis and septic shock. The team consists of infectious disease specialists, emergency physicians, and critical care doctors.

Due to the heterogeneity of such programs worldwide, it is important to assess the effectiveness of the performance improvement program at Brest University Hospital by evaluating adherence to the 2021 Surviving Sepsis Campaign (SSC) guidelines before and after its implementation.

The study will include adult patients with positive blood cultures and a positive SOFA score, or with blood cultures collected, a positive SOFA score, and sepsis/septic shock confirmed by the sepsis team at Brest University Hospital. Two periods : from 01/01/2017 to 31/12/2017 and from 01/05/2022 to 30/04/2024.

The pre- and post-implementation groups will be compared, with the primary outcome being compliance with the 2021 SSC recommendations (antibiotic therapy, hemodynamic management, respiratory support, corticosteroid therapy). Secondary outcomes include time from admission to first physician contact, time from first contact to initiation of antibiotic therapy, time from first contact to first fluid resuscitation, the proportion of sepsis patients progressing to septic shock in the emergency department, length of ICU and hospital stay, 90-day mortality, duration of mechanical ventilation, and changes in SOFA score (at 24 hours, Day 2, and Day 7).

The role of the Initial Orientation Nurse (ION) is integrated into the evaluation criteria. Using a triage grid, sometimes in collaboration with the senior emergency physician or resuscitation physician, the ION determines the optimal time frame for care and the most appropriate treatment pathway. The ION plays a key role in the early recognition of sepsis/septic shock.

The investigators will consider the time from patient evaluation by the ION to assess the speed of activation of the appropriate care pathway and the promptness of sepsis/septic shock management after recognition.

The objective of this study is to evaluate the impact of implementing a performance improvement program on the initial management of sepsis and septic shock in adults in the emergency medicine department of Brest University Hospital, guided by the 2021 Surviving Sepsis Campaign (SSC) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Major
* Patients with positive blood cultures and a positive SOFA score
* Patients with blood cultures collected, a positive SOFA score, and sepsis/septic shock confirmed by the sepsis team at Brest University Hospital.
* Patients enrolled in a social security scheme

Exclusion Criteria:

* Patients under judicial protection (guardianship, curatorship, etc.)
* Refusal to participate
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with blood cultures collected and a SOFA score ≥ 2 presenting to the emergency department of Brest University Hospital, between January 1, 2017, to December 31, 2017 and May 1, 2022, to April 30, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Delay from Initial Orientation Nurse (ION) to initiation of antibiotic therapy | Up to 6 hours
  Delay from Initial Orientation Nurse (ION) to initiation of antibiotic therapy in minutes.
  From ION assessment to the first antibiotic administration in the emergency departement.

SECONDARY OUTCOMES:
Quality of selected antibiotic therapy | Up to 6hours
  The investigators use modified Gyssen score to evaluate the quality of antibiotic therapy.
  It's a qualitative score; the response is whether the antibiotic is adapted or not.
  At the time of the administration of the first dose of antibiotic in the emergency departement.
Delay from Initial Orientation Nurse (ION) to initial fluid resuscitation | Up to 6 hours
  Delay from Initial Orientation Nurse (ION) to initial fluid resuscitation in minutes.
  From ION assessment to the first fluid administration in the emergency departement.
Quality of fluid resuscitation | Up to 3 hours
  Quality of fluid resuscitation is defined as a minimum of 30 mL/kg within 3 hours using crystalloid solutions, with a target mean arterial pressure (MAP) of 65 mmHg.
  From ION assessment, to 3hours in the emergency departement.
Quality of oxygen therapy | Up to 6 hours
  Quality of oxygen therapy is defined as maintaining an SpO2 target of 94-96%, or 88-92% if the patient has chronic respiratory failure.
  At the ION, at 3 hours, and at 6 hours in the emergency department.
Proportion of sepsis patients progressing to septic shock in the emergency department | Up to 6 hours
  Progression of sepsis to septic shock is defined by the necessity for the administration of vasopressors to achieve a mean arterial pressure (MAP) of 65 mmHg after 3 hours in the emergency department.
Duration of hospitalization in the ICU and hospital, and length of stay in the emergency department | Through study completion, an average of 6 months
  Duration of hospitalization in the ICU and hospital in days; and length of stay in the emergency department in hours.
Duration of mechanical ventilation | Through study completion, an average of 6 months
  Duration of mechanical ventilation is defined as the cumulative time of intubation (IOT) with invasive ventilation (IV) in days during hospitalization in the ICU following initial care in emergency departement.
Changes in the SOFA score | Up to day 7
  Calculation of the SOFA score. At ION in emergency departement, 24 hours, Day 2, and Day 7. The SOFA score is out of 24, and it is considered positive from 2 points onwards. The higher the score, the greater the severity.
28-day mortality | Up to days 28
  Death within 28 days of administrative admission.
90-day mortality | Up to days 90
  Death within 90 days of administrative admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement

REFERENCES:
- [Background] Rezig S, Branthome S, Basset A, Helies R, Fiore C, Bailly P, et al. Une "Sepsis Team" est elle indispensable dans chaque hopital ? Médecine Mal Infect. 1 juin 2019;49:S55-6.
- [Background] Rudd KE, Johnson SC, Agesa KM, Shackelford KA, Tsoi D, Kievlan DR, Colombara DV, Ikuta KS, Kissoon N, Finfer S, Fleischmann-Struzek C, Machado FR, Reinhart KK, Rowan K, Seymour CW, Watson RS, West TE, Marinho F, Hay SI, Lozano R, Lopez AD, Angus DC, Murray CJL, Naghavi M. Global, regional, and national sepsis incidence and mortality, 1990-2017: analysis for the Global Burden of Disease Study. Lancet. 2020 Jan 18;395(10219):200-211. doi: 10.1016/S0140-6736(19)32989-7. PMID 31954465
- [Background] Damiani E, Donati A, Serafini G, Rinaldi L, Adrario E, Pelaia P, Busani S, Girardis M. Effect of performance improvement programs on compliance with sepsis bundles and mortality: a systematic review and meta-analysis of observational studies. PLoS One. 2015 May 6;10(5):e0125827. doi: 10.1371/journal.pone.0125827. eCollection 2015. PMID 25946168
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Hylander Moller M, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock 2021. Crit Care Med. 2021 Nov 1;49(11):e1063-e1143. doi: 10.1097/CCM.0000000000005337. No abstract available. PMID 34605781
- [Background] Chiu C, Legrand M. Epidemiology of sepsis and septic shock. Curr Opin Anaesthesiol. 2021 Apr 1;34(2):71-76. doi: 10.1097/ACO.0000000000000958. PMID 33492864
- [Background] Schinkel M, Holleman F, Vleghels R, Brugman K, Ridderikhof ML, Dzelili M, Nanayakkara PWB, Wiersinga WJ. The impact of a sepsis performance improvement program in the emergency department: a before-after intervention study. Infection. 2023 Aug;51(4):945-954. doi: 10.1007/s15010-022-01957-x. Epub 2022 Nov 17. PMID 36394818